CLINICAL TRIAL: NCT00463723
Title: Topical FK506 (Tacrolimus) for Prevention of Immune Reactions Following Penetrating Keratoplasty
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FR-2000-2003
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 1999-08

CONDITIONS: Penetrating Keratoplasty
Keywords: penetrating keratoplasty; graft rejection; immunosuppression
MeSH Terms: interventions — Tacrolimus; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: FK506 0.06% (eye drops)

SUMMARY:
Background: Patients following allogeneic keratoplasty are treated with topical and frequently with systemic steroids to prevent immune reactions. Steroids are known to yield good results, but exert a wide range of side effects. The efficacy of topial FK506 in preventing immune reactions has already been demonstrated experimentally. FK506, an IL-2-inhibitor like Cyclosporin A (CSA), is known to be approximately 100 fold more potent than CSA. Aim of the study: In this study the efficacy and safety of topical FK506 will be compared to our standard treatment (i.e. steroids) after penetrating normal-risk keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Penetrating keratoplasty for Keratoconus
* Penetrating keratoplasty for Fuchs endothelial dystrophie
* Penetrating keratoplasty for Bullous keratopathy

Exclusion Criteria:

* Glaucoma
* Limbal stem cell deficiency
* Herpetic eye disease
* Repeat Keratoplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reinhard, MD, Study Chair — University eye hospital Freiburg, Germany

REFERENCES:
- [Result] Reinhard T, Mayweg S, Reis A, Sundmacher R. Topical FK506 as immunoprophylaxis after allogeneic penetrating normal-risk keratoplasty: a randomized clinical pilot study. Transpl Int. 2005 Feb;18(2):193-7. doi: 10.1111/j.1432-2277.2004.00006.x. PMID 15691272